CLINICAL TRIAL: NCT02061189
Title: Physical Exercise and Neuromuscular Diseases: Pilot Study of an Innovative Physiotherapy in Patients With Infantile Spinal Muscular Atrophy
Brief Title: Pilot Study of an Innovative Physiotherapy in Patients With Infantile Spinal Muscular Atrophy (SMA)
Acronym: ExerASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120124; 2013-A01331-44 (Other: IDRCB)
Record Dates: First submitted 2014-01-10; First posted 2014-02-12 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Infantile Spinal Muscular Atrophy of Type 2 or 3
Keywords: neuromuscular disease, Spinal Muscular Atrophy, Infantile,; motor function measure, Hammersmith scale,; rehabilitation program, physical exercise
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Atrophy, Spinal; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Swimming pool training group (Experimental): 10 patients will be selected to perform a 6 months training in a swimming pool, from M12 to M18 or M18 to M24 or M24 to M36, in defined and reproducible conditions.
  * M0, M6, M12 and M18 or M0, M6, M12, M18 and M24 or M0, M6, M12, M18, M24 and M30 assessments: Medical examination + MFM + Hammersmith scale + Non-invasive motor capacity analysis.
  * M12 to M18 or M18 to M24 or M24 to M30: Physical exercise in a swimming pool (3 times per week).
  * M24 or M30 or M36: Medical examination + MFM + Hammersmith scale + Non-invasive motor capacity analysis.
  Interventions: Other: Physical exercise in a swimming pool during 6 months
- Control group (No Intervention): 20 patients with same assessments at M0, M6, M12 and M18, but:
  * without swimming pool training.
  * without M24 assessment.

INTERVENTIONS:
Other: Physical exercise in a swimming pool during 6 months — 10 patients will undergo a training program of physical exercise in a swimming pool, 3 days per week during 6 months. Each session will last for 20 minutes.
  Arms: Swimming pool training group

SUMMARY:
This clinical trial aims to test a new physio-therapeutic approach tailored to type 2 and 3 Spinal Muscular Atrophy patients, based on physical training in swimming-pool. This specific exercise should promote motor skills of trained patients, as we have observed in different mouse models. Patient's motor skills will be assessed using different scales including MFM and Hammersmith.

This clinical trial attempts to develop a new non-invasive motor scale with sophisticated instruments.

This scale will be useful in future clinical trials on SMA, given the lack of sensitivity of currently available scales.

In addition, the study attempts to validate a questionnaire on post-exercise physical well-being.

DETAILED DESCRIPTION:
This multicenter study is based on a longitudinal assessment of the natural disease progression and on the effects of exercise protocol in a swimming pool. This study will compare patients to themselves after determining motor skills and the disease natural course for 12 months.

The study will compare different scales (MFM, Hammersmith) to our new innovative scale based on non-invasive analysis of motor skills.

30 patients will be enrolled and tested with MFM, Hammersmith and our non-invasive scale every 6 months for a total of 18 to 36 months due to the slow natural progression of the disease.

Among these 30 patients, 10 patients will be selected to perform a 6 months training in a swimming pool, from 12 to 18 months or 18 to 24 months or 24 to 30 months after enrollment, in defined and reproducible conditions.

These trained patients will finally be reassessed at 18 and 24 months or 24 and 30 months or 30 and 36 months to test the therapeutic effect of the training compared to the slope of the natural disease progression, and other parameters.

Only patients who have undergone training in the swimming pool will be reevaluated at 24 or 30 or 36 months (6 months post-training) to assess long term exercise effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with type II SMA who can sustain a sitting position without orthopedic corset or type III SMA, with genetic confirmation of the disease.
2. Age from 5 to 10 years old.
3. Patient able to understand and execute training instructions, and perform predetermined movements.
4. Patient able to achieve physical exercises in a swimming pool.
5. MFM score > 35.
6. Patient having any contraindication to physical rehabilitation in a swimming pool.
7. Consent signed by the holders of parental responsibility for children participating in the study.
8. Patient with social security insurance.

Exclusion Criteria:

1. Pneumonia: the inclusion is to be delayed for at least 3 months after recovery of infection.
2. Heart, renal or hepatic failure.
3. Patient undergoing a major surgery during the study: spinal fusion.
4. Patient under the care of a guardian.
5. Inability to cooperate.
6. Medication potentially interfering with the SMA (i.e., riluzole, salbutamol, phenylbutyrate, sodium valproate) started less than 6 months before inclusion.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Motor function measurement (MFM) | 18 months (control group) to 36 months maximum (swimming pool group)
  The motor ability of all patients will be followed for 18 or 24 months, for a total of four or five functional assessments, 1 every 6 months. Each patient will be assessed with the MFM.

SECONDARY OUTCOMES:
Hammersmith scale | M18 or M24 or M30 or M36
  Motor Assessments will be performed in the same order : MFM first, then Hammersmith scale.
Questionnaire on post-exercise physical well-being | M18 or M24 or M30 or M36
  Force and pain felt assessment by questionnaire just before and after each physical training session for 6 months.
Non invasive motor capacity assessment | M18 or M24 or M30 or M36
  Monitoring motor capacity with a non-invasive sophisticated instrument operating in the Paris Descartes University platform. This monitoring will be performed for 18 or 24 months, for a total of four or five functional assessments, 1 every 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Susana QUIJANO-ROY, MD, PhD, Principal Investigator — Raymond Poincaré Hospital, Garches, FRANCE
Locations (1):
- Raymond Poincaré Hospital, Garches, Hauts-de-Seine, France